CLINICAL TRIAL: NCT02229786
Title: Buscopan® Plus, Buscopan®, Paracetamol and Placebo: Double-blind Randomized Group Comparison to Investigate the Efficacy and Tolerability of the Film-coated Tablets in Patients With Painful Gastric or Intestinal Spasms
Brief Title: Efficacy and Tolerability of Buscopan Plus in Painful Gastric or Intestinal Spasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218.202
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Butylscopolammonium Bromide; Acetaminophen

ARMS (4):
- Buscopan® plus (Experimental)
  Interventions: Drug: Buscopan® plus
- Buscopan® (Active Comparator)
  Interventions: Drug: Buscopan®
- Paracetamol (Active Comparator)
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buscopan® plus
  Arms: Buscopan® plus
Drug: Buscopan®
  Arms: Buscopan®
Drug: Paracetamol
  Arms: Paracetamol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate efficacy and tolerability of Buscopan® plus versus Buscopan®, paracetamol, and placebo in patients with painful gastric or intestinal spasms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age: 18 - 70 years
* Diagnosis: recurring painful gastric or intestinal spasms such as occur e.g. in irritable bowel syndrome, which are not organic in origin, have been present for at least 2 months, and are serious enough to interfere with everyday activities
* Patient briefing as per §§ 40/41 of the Arzneimittelgesetz (AMG) and patient's declaration of Informed Consent in writing, in agreement with Good Clinical Practice (GCP) and current legal requirements
* A pain assessment of 3 cm or more on the visual analog scale on at least one of the 2 days immediately preceding the second visit

Exclusion Criteria:

* Painful gastric or intestinal spasms of organic origin such as Crohn's disease, ulcerative colitis, lactose intolerance
* Tumour pain/malignant growths
* Patients with other severe pain states of organic origin (e.g. biliary colic)
* Mechanical stenoses of the gastrointestinal tract, megacolon
* Urinary retention associated with mechanical stenoses of the urinary tract (e.g. in prostate adenoma)
* Narrow-angle glaucoma
* Tachyarrhythmia
* Myasthenia gravis
* Glucose 6-phosphate dehydrogenase deficiency (danger of haemolytic anaemia)
* Known hypersensitivity to N-butylscopolammonium bromide or paracetamol
* Severe liver impairment (e.g. through chronic alcohol abuse, hepatitis):

  * a) Serum-Glutamate-Oxalacetat-Transaminase/ Aspartate Aminotransferase (SGOT) higher than four times the norm
  * b) Bilirubin > 3 mg/dl
  * c) Quick's value < 70%
* Meulengracht-Gilbert syndrome (metabolic disturbance with episodes of jaundice)
* Severe kidney failure: creatinine > 2 mg/dl
* Known depression or known mental illness, anxiety disturbance
* Concomitant intake of analgesics, nonsteroidal antiinflammatory drugs (NSAIDs) and/or spasmolytics, anticholinergics, nitrates
* Concomitant medication affecting gastrointestinal motility
* Regular (daily) use of laxatives
* Drugs that induce liver enzymes
* Concomitant administration of chloramphenicol
* Use of narcotics
* Antidepressant treatment or treatment with psychoactive drugs
* Pregnancy and lactation
* Alcohol abuse (more than 60 g alcohol/day)
* Frequent vomiting that might prevent adequate absorption of the active ingredient after the film-coated tablet is taken
* Patients who are unlikely to be able to keep the examination appointments or cannot reliably take the study medication regularly
* Simultaneous participation in another clinical study
* Patients who are not trained in the VAS (PI) at Visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1637 (Actual)
Dates: Start 1998-02; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Mean decrease in pain intensity on a VAS (visual analog scale) | 3 weeks

SECONDARY OUTCOMES:
Frequency of pain on a 4-stage verbal rating scale | up to 4 weeks
Global assessment of efficacy by patient on a 5-point rating scale | up to 4 weeks
Global assessment of efficacy by investigator on a 5-point rating scale | up to 4 weeks
Number of patients with adverse events | up to 4 weeks